CLINICAL TRIAL: NCT00066586
Title: A Randomized Study Of The Effect Of Exemestane (Aromasin) Versus Placebo On Breast Density In Postmenopausal Women At Increased Risk For Development Of Breast Cancer
Brief Title: Exemestane in Reducing Breast Density in Postmenopausal Women at Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MAP2; CAN-NCIC-MAP2 (Other: PDQ Identifier); PFIZER-971-ONC-0028-088 (Other: Pfizer); CDR0000316328 (Other: PDQ); NCT00258648 (obsolete NCT alias)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exemestane (Active Comparator)
  Interventions: Drug: exemestane
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: exemestane — exemestane 25 mg once daily x 1 year
  Arms: Exemestane
Drug: Placebo — placebo once daily x 1 year
  Arms: Placebo

SUMMARY:
RATIONALE: High estrogen levels may be associated with dense breast tissue and an increased risk of developing breast cancer. Exemestane may be effective in preventing the development of breast cancer by decreasing estrogen levels and reducing breast density.

PURPOSE: Randomized clinical trial to study the effectiveness of exemestane in preventing the development of breast cancer by decreasing estrogen levels and reducing breast density in postmenopausal women who are at increased risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of exemestane in decreasing breast density at least 1 grade in postmenopausal women with increased radiological breast density at increased risk for breast cancer.
* Determine whether the decrease in breast density is sustained 1 year after the cessation of this drug in these participants.
* Correlate the grade of breast density with bone density at baseline and at 1 year in participants treated with this drug.
* Determine the overall safety of this drug, in terms of bone and lipid metabolism and toxicity, in these participants.
* Determine the menopause-specific quality of life of participants treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Participants are stratified according to baseline mammographic density grade (2 vs 3 vs 4 vs 5 vs 6). Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive oral exemestane once daily for 1 year.
* Arm II: Participants receive oral placebo once daily for 1 year. In both arms, treatment continues in the absence of disease or unacceptable toxicity.

Quality of life is assessed at baseline and then at 3, 6, 9, 12, 18, and 24 months.

Participants are followed at 18 and 24 months.

PROJECTED ACCRUAL: A total of 120 participants (60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Radiologically confirmed density occupying at least 25% of the breast tissue on baseline mammogram*

  * Grade 2, 3, 4, 5, or 6 (Boyd classification)

    * Participants with different grades between the 2 breasts should be classified according to a higher grade NOTE: *Performed within 6 months before study entry
* Bone mineral density T-score of either posterior-anterior spine or hip (femoral neck) must be no greater than 2.0 standard deviations below the mean value of peak bone mass in young normal women as determined by DEXA scan within the past 6 months
* No concurrent breast cancer
* No prior invasive breast cancer or ductal carcinoma in situ
* No breast implants
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal, defined as 1 of the following:

  * Over 50 years of age with no spontaneous menses for at least 1 year
  * 50 years of age and under with no menses (e.g., spontaneous or secondary to hysterectomy) within the past year AND a follicle-stimulating hormone level within institution postmenopausal range
  * Bilateral oophorectomy

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Cardiovascular

* No cardiovascular disease
* No history of myocardial infarction
* No history of stroke
* No uncontrolled high blood pressure

Other

* No uncontrolled metabolic or endocrine disease
* No malabsorption syndrome
* No known hypersensitivity to exemestane or its excipients
* No other malignancy within the past 5 years except curatively treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy
* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* More than 3 months since prior exogenous estrogen and/or progesterone/progestin therapy
* More than 6 months since prior selective estrogen-receptor modulators (e.g., tamoxifen, toremifene, or raloxifene)
* No concurrent selective estrogen-receptor modulators (e.g., tamoxifen, toremifene, or raloxifene)
* No concurrent steroids
* Vaginal estrogens allowed (e.g., Estring® or Vagifem®)

  * No concurrent compounded creams

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 4 weeks since prior investigational agents
* No other concurrent medications that would preclude study endpoints
* No concurrent over-the-counter products or supplements considered to have an estrogenic effect, including any of the following:

  * Ginseng
  * Ginkgo biloba
  * Black cohosh
  * Dong quai
  * Fortified soy supplements (e.g., phytoestrogen preparations)

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2001-08-01 (Actual); Primary Completion 2007-11-16 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Change in breast density as measured by Boyd Scale at 1 year | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Goss, MD, PhD, Study Chair — Massachusetts General Hospital
Locations (12):
- United States (8):
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
- Canada (4):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Northwestern Ontario Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cigler T, Richardson H, Yaffe MJ, Fabian CJ, Johnston D, Ingle JN, Nassif E, Brunner RL, Wood ME, Pater JL, Hu H, Qi S, Tu D, Goss PE. A randomized, placebo-controlled trial (NCIC CTG MAP.2) examining the effects of exemestane on mammographic breast density, bone density, markers of bone metabolism and serum lipid levels in postmenopausal women. Breast Cancer Res Treat. 2011 Apr;126(2):453-61. doi: 10.1007/s10549-010-1322-0. Epub 2011 Jan 9. PMID 21221773